CLINICAL TRIAL: NCT06397170
Title: Effects of Graded Repetitive Arm Supplementary Program Versus Task Based Training on Upper Limb Function in Stroke Patients
Brief Title: Graded Repetitive Arm Supplementary Program Versus Task Based Training on Upper Limb Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0281
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Upper Extremity Paresis; Motor Activity
Keywords: Stroke; Upper Extremity Paresis; Motor Activity
MeSH Terms: conditions — Stroke; Paresis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be divided into Group A (N=19) will receive Graded repetitive arm supplementary program and Patients in Group B (N=19)will receive Task based training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded repetitive arm supplementary program group (Experimental): Patients in Group A will receive Graded repetitive arm supplementary program.
  Interventions: Other: Graded repetitive arm supplementary program
- Task based training group (Active Comparator): Patients in Group B will receive Task based training.
  Interventions: Other: Task based training

INTERVENTIONS:
Other: Graded repetitive arm supplementary program — Patients in Group A will receive Graded repetitive arm supplementary program
  Arms: Graded repetitive arm supplementary program group
Other: Task based training — Patients in Group B will receive Task based training.
  Arms: Task based training group

SUMMARY:
To determine effects of graded repetitive arm supplementary program versus Task based training on Upper limb function in stroke patients.

DETAILED DESCRIPTION:
This study will be Randomized Clinical Trial. A total of 38 stroke patients will be recruited by using non-probability convenience sampling Technique. Patients will be Randomized and allocated into two interventional groups based on the inclusion and exclusion criteria. Patients in Group A will receive Graded repetitive arm supplementary program and Patients in Group B will receive Task based training. All participants will receive the treatment for 40 minutes per session, 5 days per week for 5 weeks. For the evaluation of all participant scales like be Chedoke Arm and Hand Activity Inventory for clinical relevance, Fugl Mayer assessment scale for performance assessment, Action Reach Arm Test for coordination and dexterity and Motor Activity Log for functional assessment of Upper limb in stroke patients. D

ELIGIBILITY:
Inclusion Criteria:

* Patients with Sub acute stage of stroke.
* Patients with Ischemic and Haemorrhagic stroke.
* Patients with Cognition level on Mini Mental State Examination must be > 24
* Patients with mild pain in upper extremity according to Numeric Pain Rating Scale
* Patients with Grade 2 active movements in affected extremity Tone of upper limb at Modified Ashworth Scale Grade 1+.

Exclusion Criteria:

* Other neurological disorders e.g. brain tumor, encephalitis, meningitis, brain abscess.
* Use of antipsychotics
* Use of drugs for spasticity.
* Patients with vestibular impairment.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Fugl Mayer assessment scale | 6 months
  It is designed to assess reflex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia. total score is 126.This tool has an excellent Inter- and intrarater reliability (intra class correlation coefficient = 0.98-0.99), validity is also excellent (r = 0.74-0.93, P < .0001). Higher scores indicate maximum recovery. higher the score greater is the improvement
The Motor Activity Log (MAL) | 6 months
  The Motor Activity Log (MAL) is a subjective outcome measure of an individual's real life functional upper limb performance. The Motor activity log is administered by semi-structured interview and items are scored by patients according to their performance of each task over the past 7 days. The MAL adopts a 6-point ordinal scale, although patients can attribute a half-score, resulting in 11-point Likert scales with specified anchoring definitions at 6 points. higher the score greater is the improvement

CONTACTS AND LOCATIONS:
Overall Officials: Zeest hashmi, Principal Investigator — Riphah International University
Locations (1):
- Imran International Amjad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connell LA, McMahon NE, Watkins CL, Eng JJ. Therapists' use of the Graded Repetitive Arm Supplementary Program (GRASP) intervention: a practice implementation survey study. Phys Ther. 2014 May;94(5):632-43. doi: 10.2522/ptj.20130240. Epub 2014 Feb 6. PMID 24505098
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Yang CL, Waterson S, Eng JJ. Implementation and Evaluation of the Virtual Graded Repetitive Arm Supplementary Program (GRASP) for Individuals With Stroke During the COVID-19 Pandemic and Beyond. Phys Ther. 2021 Jun 1;101(6):pzab083. doi: 10.1093/ptj/pzab083. PMID 33682872
- [Background] Lee HS, Lim JH, Jeon BH, Song CS. Non-immersive Virtual Reality Rehabilitation Applied to a Task-oriented Approach for Stroke Patients: A Randomized Controlled Trial. Restor Neurol Neurosci. 2020;38(2):165-172. doi: 10.3233/RNN-190975. PMID 32176674